CLINICAL TRIAL: NCT00361127
Title: Influence of ACE Genotype on Lung Diffusion at Rest and After Fluid Overload in Heart Failure Patients Treated With ACE-inhibitors
Brief Title: Influence of Angiotensin Converting Enzyme (ACE) Genotype on Lung Diffusion in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piergiuseppe Agostoni (Other)
Responsible Party: Sponsor-Investigator, Piergiuseppe Agostoni, MD PhD, Centro Cardiologico Monzino
Organization: Centro Cardiologico Monzino (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCM S65/206
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure, Congestive
Keywords: Heart failure; pulmonary edema; ACE-inhibitors; lung diffusion; exercise capacity; Chronic heart failure
MeSH Terms: conditions — Heart Failure; Pulmonary Edema

ARMS (1):
- CMPD patients (Experimental): Patients with CMPD with evaluation of ACE I/D polymorphism
  Interventions: Drug: isotonic saline infusion

INTERVENTIONS:
Drug: isotonic saline infusion

SUMMARY:
In patients with chronic heart failure ACE-inhibitor treatment improves lung diffusion and prevents pulmonary edema after fluid overload. In the western country, 3 population types of ACE genotypes exist (DD, ID, II). It is unknown whether the ACE genotype influences the response to fluid overload in ACE-inhibitor treated chronic heart failure patients.

DETAILED DESCRIPTION:
Patients with chronic heart failure in stable clinical condition treated with ACE-inhibitors, but not aspirin, will be evaluated by means of maximal cardiopulmonary exercise test and lung function including lung diffusion measurements. These tests will be done before and after rapid 500 ml isotonic saline infusion. Patients will be grouped according to their ACE genotype.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) class I and II heart failure
* Chronic ACE-inhibitor treatment

Exclusion Criteria:

* Aspirin treatment in the previous 2 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Possible identification of a genetic pattern responsible for different responses to ACE-inhibition during fluid overload in heart failure | Third day

SECONDARY OUTCOMES:
Influence of ACE-genotype on exercise capacity | Third day
Influence of ACE-genotype on lung function | Third day

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, MD.PhD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy

REFERENCES:
- [Background] Agostoni P, Cattadori G, Bianchi M, Wasserman K. Exercise-induced pulmonary edema in heart failure. Circulation. 2003 Nov 25;108(21):2666-71. doi: 10.1161/01.CIR.0000097115.61309.59. Epub 2003 Oct 27. PMID 14581402
- [Background] Guazzi M, Marenzi G, Alimento M, Contini M, Agostoni P. Improvement of alveolar-capillary membrane diffusing capacity with enalapril in chronic heart failure and counteracting effect of aspirin. Circulation. 1997 Apr 1;95(7):1930-6. doi: 10.1161/01.cir.95.7.1930. PMID 9107182